CLINICAL TRIAL: NCT00348842
Title: Phase II: Safety and Primary Efficacy of Clinical Application of Newcastle Disease Virus for the Treatment of Patients Resistant to All Conventional Modalities
Brief Title: Newcastle Disease Virus (NDV) for Cancer Patients Resistant to Conventional Anti-cancer Modalities
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 397231205-HMO-CTIL
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2006-02

CONDITIONS: Metastatic Cancer; Newcastle Disease Virus (NDV)
Keywords: Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis

INTERVENTIONS:
Procedure: Newcastle Virus

SUMMARY:
NDV is a virus tht is harmful in chicken, but harmless in man. There are 2 major sub-strains of NDV, one oncolytic and one non-oncolytic. Oncolytic NDV (MTH-68H) preferentially homes and replicates in cancer cells and therefore, administration of NDV intravenously or preferentially intra-tumor, either by direct injection or by injection into an afferent artery results in direct lysis of tumor cells. NDV activates apoptotic mechanism in cancer cells and thus, results in natural cell death.

Both oncolytic and non-oncolytic NDV were used clinically in hundreds of patients with different types of cancer worldwide. NDV were proved harmless in man. Clinical studies were done for more than a decade and the efficacy of NDV was documented on pre-clinical animals models as well as in man.

For a large number of patients with metastatic cancer and chemotherapy resistant hematological malignances, no cure can be provided by conventional anti-cancer modalities, new treatment options are urgently indicated. The goal of the study is to use NDV, in order to provide such treatment for patients in need.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following disease category will be eligible:

Patients with metastatic lung cancer, metastatic GI cancer, metastatic urogenital cancer, skin and soft tissue cancer.

* Failure to anti-cancer modalties and evidence of progressive disease despite optimal application of all relevant available anti-cancer modalities.
* Consenting patients.
* The patient should sign a consent form stating that he/she will make sure to avoid any contact with chicken or any other species of birds.

Exclusion Criteria:

* Not fulfilling any of the above criteria.
* Moribund patients or patients with life-expectancy <3 months.
* Karnofsky performance status <60%.
* Pregnant or lactating women.
* Active local or systemic infections requiring treatment.
* Co-morbidity or life-threatening clinical condtion other than the basic cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-03; Study Completion 2006-06 (Estimated)

PRIMARY OUTCOMES:
Safety and primary efficacy of NDV treatment in cancer patients who failed conventional modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel